CLINICAL TRIAL: NCT04176185
Title: A Phase III Trial Evaluating the Efficacy and Safety of the House Dust Mite (HDM) Sublingual Immunotherapy (SLIT)-Tablet in Adult Chinese Subjects With HDM Allergic Rhinitis/Rhinoconjunctivitis Using an Environmental Exposure Chamber
Brief Title: A Research Study in Chinese People With Allergy to House Dust Mites, Using an Environmental Exposure Chamber
Acronym: QUEST
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: COVID-19
Sponsor: ALK-Abelló A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MT-16
Record Dates: First submitted 2019-10-25; First posted 2019-11-25 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2021-02

CONDITIONS: Allergic Rhinoconjunctivitis
Keywords: House Dust Mite; Allergic rhinitis; Allergic conjunctivitis; China; Environmental exposure chamber
MeSH Terms: conditions — Rhinitis, Allergic; Conjunctivitis, Allergic

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Investigator
Masking Description: Randomised
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Experimental): HDM SLIT-tablet once daily for approximately 24 weeks
  Interventions: Biological: Sublingual allergy immunological tablet
- Placebo (Placebo Comparator): Placebo tablet once daily for approximately 24 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Sublingual allergy immunological tablet — For daily administration (1 tablet per day)
  Other Names: 12 SQ HDM SLIT-tablet; Acarizax
  Arms: Active
Other: Placebo — For daily administration (1 tablet per day)
  Other Names: Placebo sublingual tablet
  Arms: Placebo

SUMMARY:
This trial evaluates the efficacy and safety of HDM SLIT-tablet in treatment of HDM AR. The efficacy is evaluated using an environmental exposure chamber (EEC). Subjects will be randomised to receive treatment with HDM SLIT-tablet and placebo 1:1.

DETAILED DESCRIPTION:
This trial is a 24 weeks, randomised, parallel-group, double-blind, placebo-controlled phase III trial. Approximately 202 subjects will be randomised (1:1) to receive treatment with HDM SLIT-tablet or placebo. The trial will be conducted in China, with subjects recruited and treated in China. Two EEC assessments (baseline and end of treatment) will take place at a validated EEC facility in Austria.

The primary objective is to demonstrate the efficacy of the HDM SLIT-tablet (12 SQ-HDM) once daily compared to placebo in the treatment of HDM AR nasal symptom determined during the EEC session at week 24.

ELIGIBILITY:
Inclusion criteria

* Male or female Chinese subjects aged ≥18 years
* A clinical history of HDM AR/C with or without asthma
* Positive SPT and IgE to Der p or Der f at screening
* A TNSS of at least 6 of 12 within the first 2 hours of the screening EEC session prior to randomisation

Exclusion criteria

* Sensitised and regularly exposed perennial or seasonal allergens
* Asthma requiring treatment with high-dose ICS
* Reduced lung function
* Has a nasal condition that could confound the efficacy or safety assessment
* A relevant history of systemic allergic reaction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2019-12-17 (Actual); Study Completion 2022-01-19 (Actual)

PRIMARY OUTCOMES:
Total Nasal Symptom Score (TNSS) | Last 4 hours of the EEC session at week 24
  Primary endpoint, average TNSS during the EEC session at week 24, defined as the average of all TNSS observed in the last 4 hours of the EEC session at week 24. Measured on a scale of 0 (no symptoms) to 12 (severe symptoms).

SECONDARY OUTCOMES:
Total Symptom Score (TSS) | Last 4 hours of the EEC session at week 24
  Key secondary endpoint, average TSS during the EEC session at week 24, defined as the sum of the Total Ocular Symptom Score (TOSS) and TNSS observed in the last 4 hours of the EEC session at week 24. Measured on a scale of 0 (no symptoms) to 18 (severe symptoms).

OTHER OUTCOMES:
Frequency of adverse events | 26 weeks
  Number of Adverse events per treatment group
Assessment of lung function | 26 weeks
  FEV1
Total Ocular Symptom Score (TOSS) | Last 4 hours of the EEC session at week 24
  Average TOSS during the EEC session at week 24, defined as the average of all TOSS observed in the last 4 hours of the EEC session at week 24. Measured on a scale of 0 (no symptoms) to 6 (severe symptoms).
Immunology | Baseline to 24 weeks
  Change from baseline in measurements of house-dust-mite-specific IgG & IgE antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Luo Zhang, Prof., Principal Investigator — Beijing Tongren Hospital
Locations (2):
- Vienna Challenge Chamber, Vienna, Austria
- Tongren Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No